CLINICAL TRIAL: NCT01657786
Title: Association of 5-HT3 Receptor Gene Polymorphism With the Efficiency of Ondansetron for Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 4-2008-0075
Record Dates: First submitted 2012-07-28; First posted 2012-08-06 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Post Operative Nausea and Vomiting
Keywords: ondanstron; gene polymorphism; postoperative nausea and vomiting; laparoscopic surgery under general anesthesia
MeSH Terms: conditions — Vomiting; Postoperative Nausea and Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ondansetron administration group (Experimental)
  Interventions: Dietary Supplement: administration of ondanstron and screening of genomic DNA

INTERVENTIONS:
Dietary Supplement: administration of ondanstron and screening of genomic DNA — Thirty minutes before the end of surgery, ondansetron 0.1 mg/kg is administered intravenously. We assess an episode of PONV at first 2 h and 2-24 h after surgery. Genomic DNA was prepared and screened. The incidence of PONV is compared among genotypes in 5-HT3 receptor gene polymorphisms (5-HT3a: S253N; 5-HT3b: Y129S, -100_-102delAAG).

SUMMARY:
Postoperative nausea and vomiting (PONV) is a common and distressing complication in patients undergoing general anesthesia. However, although 5-hydroxytryptamine type 3 (5-HT3) receptor antagonists have significantly reduced PONV, it is reported that over 35% of patients treated with ondansetron experience PONV. Though the cause of failure in ondansetron treatment is not clear, the investigators assumed that polymorphism in the 5-HT3 receptor gene would contribute to such inter-individual variation. In this study, the investigators examine whether the polymorphisms of 5-HT3 receptor gene affect the efficacy of ondansetron to prevent PONV in patients undergoing general anesthesia for laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (20-90 years of age) scheduled for undergoing laparoscopic surgery undergoing general anesthesia

Exclusion Criteria:

* Patients with previous history of drug allergy,
* administration of antiemetic drugs within 24 hours,
* nausea/vomiting within 24 hours and liver or kidney disease

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2008-05; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The relationship between the incidence of PONV after ondansetron administration and genotypes in 5-HT3 receptor gene polymorphisms ((5-HT3a: S253N; 5-HT3b: Y129S, -100_-102delAAG) | at first 2 h and 2-24 h after surgery.
  The incidence of PONV after ondansetron administration is compared among genotypes in 5-HT3 receptor gene polymorphisms (5-HT3a: S253N; 5-HT3b: Y129S, -100_-102delAAG).

CONTACTS AND LOCATIONS:
Locations (1):
- Associate Professor Department of Anesthesiology and Pain Medicine, Seoul, Seoul, South Korea